CLINICAL TRIAL: NCT05469672
Title: The Effect of Low-level Laser Versus High-intensity Laser Therapy in the Management of Adhesive Capsulitis: a Randomized Clinical Trial
Brief Title: The Effect of Laser Therapy in the Management of Adhesive Capsulitis: a Randomized Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Banu Ordahan, Clinical Professor, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BOrdahan
Record Dates: First submitted 2022-07-18; First posted 2022-07-22 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Pain Disorder; Low Level Laser Therapy
Keywords: Adhesive capsulitis Pain; High-intensity laser therapy; Low-level laser therapy; Pain
MeSH Terms: conditions — Somatoform Disorders; Pain | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low-level laser therapy (Active Comparator): LLLT will be performed 3 times a week for a period of 3 weeks
  Interventions: Other: Low-level laser therapy; Other: High-intensity laser therapy
- high-intensity laser therapy (Active Comparator): HILT will be performed 3 times a week for a period of 3 weeks
  Interventions: Other: Low-level laser therapy; Other: High-intensity laser therapy

INTERVENTIONS:
Other: Low-level laser therapy — For LLLT, laser treatment will be applied using gallium-aluminum-arsenide (GaAIAs, infrared laser) diode laser (Chattanooga, Mexico, USA) at a wavelength of 904 nm, output power of 240 Mw and a frequency of 5000 Hz. The spot area is about 0.5 cm2. A total of 9 points will irradiated along the glenohumeral joint, with a power density of 3 j/cm2 at each point. The application time was 50 seconds to each point. The total dose per shoulder was 27 J per treatment. Three sessions of LILT therapy per week will administered over a three-week period.
Other: High-intensity laser therapy — HILT: A hot laser derived from a Nd: YAG laser has 12 W (watt) and 1064 nm characteristics. The device will administered to the shoulder area in two steps in the HILT group: phase I and phase II. The application will made utilizing continuous circular movements in both phases I and II. The first three sessions consisted of a 75-second intermittent phase analgesic effect at 8 W and 10 J/cm2 for a total energy of 100 J. The following six sessions consisted of a continuous 30-second bio stimulating effect with a dosage of 12 W 120 J/cm2. Over the course of three weeks, nine treatment sessions of HILT will be given.

SUMMARY:
In this study, it was aimed to compare the effects of low-level laser therapy (LLLT) and high-intensity laser therapy (HILT) on shoulder joint range of motion, level of pain and functional status in patients with adhesive capsulitis

DETAILED DESCRIPTION:
This study will be designed as a randomized, prospective, single-blind clinical trial with a 3-week follow-up. A total of 50 patients who applied to our hospital with the complaint of shoulder pain will be evaluated for inclusion in the study. Patients will be randomized into two groups as high-intensity laser (HILT) + stretching exercise group and low-level laser (LLLT) + stretching exercise group.

ELIGIBILITY:
Inclusion Criteria:

1. patients aged between 25-65 years
2. patients clinically diagnosed with adhesive capsulitis, characterized by limitation of passive external rotation of the affected shoulder to less than 50% of the contralateral shoulder and normal radiographic finding of the affected shoulder
3. patients with severe pain and shoulder limitation for at least 3 months
4. patients who are literate and able to understand verbal instructions in our language.

Exclusion Criteria:

1. Calcific tendinopathy, glenohumeral osteoarthritis, fracture, shoulder surgery, shoulder trauma, history of malignancy and infection, history of inflammatory rheumatic diseases
2. History of bilateral simultaneous adhesive capsulitis
3. Recent history of lung, breast, or bypass surgery/radiotherapy
4. History of corticosteroid injection to the same shoulder in the last 1 year
5. History of cervical radiculopathy/brachial plexus lesion
6. Neuromuscular disease history
7. History of physical therapy program for the same shoulder in the last 6 months.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-09-25 (Estimated); Primary Completion 2022-09-25 (Estimated); Study Completion 2022-10-25 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) is used to measure and monitor the intensity of pain. Change from baseline in pain on the VAS at week 3 | Baseline-Week 3
  This is a 10 cm ruler that describes painlessness at one end and the most severe pain at the other. A patient scores his/her pain from 0 to 10.

SECONDARY OUTCOMES:
Shoulder Pain and Disability Index | Baseline and week 3
  The severity of pain and limitation experienced by individuals during certain activities will be evaluated with the Shoulder Pain and Disability Index (SPADI). SPADI is an evaluation method filled by the individual, lasting approximately 5-10 minutes, which questions the state of pain and disability in the shoulder. [11] SPADI consists of 2 sections and 13 sub-headings, namely pain and disability. The first part consists of 5 questions which evaluate the worst pain level being experienced in the last 14 days, lying on the affected side, and level of pain during reaching up, reaching behind the neck, and pushing activity. The second part evaluates the disability level by questioning the level of limitation experienced by the individual during personal care, dressing and carrying activities. The total score range in the scale ranges from 0 to 130.
  Change from baseline in pain and disability on the Shoulder Pain and Disability Index at week 3
Measuring the range of motion at shoulder joint | Baseline and week 3
  Shoulder active range of motion (flexion, abduction, internal and external rotation) will be measured with a universal goniometry.
  Change from baseline in shoulder joint on the measuring the range of motion at shoulder joint at week 3

CONTACTS AND LOCATIONS:
Overall Officials: BANU ORDAHAN, Principal Investigator — Meram Medical School, Necmettin Erbakan University, Konya, Turkey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ordahan B, Yigit F, Mulkoglu C. Efficacy of Low-level Laser Versus High-intensity Laser Therapy in the Management of Adhesive Capsulitis: A Randomized Clinical Trial. Saudi J Med Med Sci. 2023 Jul-Sep;11(3):201-207. doi: 10.4103/sjmms.sjmms_626_22. Epub 2023 Jul 15. PMID 37533657